CLINICAL TRIAL: NCT07142577
Title: The Effect of Mandala Coloring on Mental Well-Being and Life Satisfaction in Elderly Individuals in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Hatice YAĞCI KARAMANLI, Principal Investigator,, Karamanoğlu Mehmetbey University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: E-67796128-819-2500015361
Record Dates: First submitted 2025-08-07; First posted 2025-08-26 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Mandala Coloring; Mental Well-being; Life Satisfaction
Keywords: life satisfaction; mental well-being; mandala coloring
MeSH Terms: conditions — Psychological Well-Being; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: It is a quasi-experimental study that includes only the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deney (Experimental): A group staying at a nursing home who will paint mandalas
  Interventions: Other: Mandala coloring

INTERVENTIONS:
Other: Mandala coloring — Mandala coloring activities will be carried out by the certified researcher 1 days (1-1,5 hours) a week for 8 weeks.

SUMMARY:
This study investigates whether mandala coloring affects life satisfaction and mental well-being in older adults. Data will be collected at the Hatice Hakkı Polat Nursing Home Elderly Care and Rehabilitation Center between September 15, 2025, and November 7, 2025. The full study will be completed in November 2025.

DETAILED DESCRIPTION:
Participation in the study is voluntary. All individuals living in a nursing home who volunteered to participate were included in the study. All elderly individuals with sufficient physical and mental capacity were contacted.

All individuals living in a nursing home who met the study criteria were included in the study group. Participants were asked to color mandalas for eight weeks. Data collection forms were administered before and after the study. Due to the current conditions at the nursing home, all participants were willing to participate in the coloring activity, and this request could not be denied. Therefore, there was no control group.

The scales will be completed face-to-face. The data obtained will be processed using SPSS. The statistical analyst will not know which group is the experimental group and which is the control group.

The results were compared before and after.

ELIGIBILITY:
Inclusion Criteria:

* Being over 65
* Residing in a nursing home
* Voluntarily participating in the study

Exclusion Criteria:

* Having a physical or mental disability that would prevent participation in the study
* Not wanting to participate in the study.

Min Age: 65 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Life satisfaction scale | 8 weeks
  The possible score on the scale ranges from 5 to 25. In the reference article, the consistency coefficient for the entire scale was calculated as r = 0.88. A higher score indicates higher life satisfaction.
Warwick-Edinburgh Mental Well-Being Scale | 8 weeks
  The scale consists of 14 items and addresses individuals' positive mental health by encompassing both psychological and subjective well-being. The Cronbach's alpha coefficient was found to be 0.89 in the reference article. As the score increases, so does the level of mental well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice YAĞCI KARAMANLI, Principal Investigator — KARAMANOĞLU MEHMETBEY UNİVERSTY
Locations (1):
- Hatice Hakkı Polat Nursing Home Elderly Care and Rehabilitation Center, Karaman, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Consent was not obtained from all co-authors.